CLINICAL TRIAL: NCT06358573
Title: Intratumoral INT230-6 Followed by Neoadjuvant Immuno-chemotherapy in Patients With Early Triple-negative Breast Cancer (TNBC). An Open-label Randomized Two-cohort Phase 2 Clinical Trial. INVINCIBLE-4-SAKK
Brief Title: Intratumoral INT230-6 Followed by Neoadjuvant Immuno-chemotherapy in Patients With Early TNBC. INVINCIBLE-4-SAKK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 66/22
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Triple-negative Breast Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: triple-negative breast cancer; TNBC; Intratumoral INT230-6; neoadjuvant immuno-chemotherapy; INT230-6; early stage
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized, open-label multicenter phase 2 clinical study to determine the clinical activity, safety and tolerability of INT230-6 in patients with early stage, operable TNBC who undergo neoadjuvant systemic treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A experimental (Experimental): Intervention 1-2 weeks:
  - 2 Injections of INT230-6 into primary tumor of the breast
  Thereafter
  * Standard of Care including surgery (30 weeks)
  * Immuno-chemotherapy -> 24 weeks
  Neoadjuvant therapy as Keynote-522 (Standard of Care) - 24 Weeks
  Pembrolizumab q3W in combination with
  * Cycles 1-4: Paclitaxel q1W + Carboplating q1W or q3W
  * Cycle 5-8: Doxorubicin or Epirubicin q3W + Cyclophospahmide q3W
  * MRI
  * Surgery
  Interventions: Drug: INT230-6; Other: neoadjuvant immuno-chemotherapy
- Cohort B Standard of Care (Other): Intervention 1-2 weeks:
  - No intervention - start of immune-chemotherapy after randomization
  Thereafter
  * Standard of Care including surgery (30 weeks)
  * Immuno-chemotherapy -> 24 weeks
  Neoadjuvant therapy as Keynote-522 (Standard of Care) - 24 Weeks
  Pembrolizumab q3W in combination with
  * Cycles 1-4: Paclitaxel q1W + Carboplating q1W or q3W
  * Cycle 5-8: Doxorubicin or Epirubicin q3W + Cyclophospahmide q3W
  * MRI
  * Surgery
  Interventions: Other: neoadjuvant immuno-chemotherapy

INTERVENTIONS:
Drug: INT230-6 — INT230-6 is a formulation consisting of an proprietary amphiphilic cell penetration enhancer molecule, 8-((2-hydroxybenzoyl)amino)octanoate, also referred to as SHAO, combined with cisplatin and vinblastine sulfate.
  The IMP is without marketing authorization in Switzerland and anywhere in the world.
  Arms: Cohort A experimental
Other: neoadjuvant immuno-chemotherapy — Standard of care

SUMMARY:
About 10-20% of all individuals with breast cancer have a so-called triple-negative tumor (TNBC). This type of breast cancer has a particularly unfavorable course and a higher mortality rate compared to other forms of breast cancer. Research studies show that it is important for individuals with TNBC to achieve a so-called pathologic complete response (pCR) to treatment. In the phase II study SAKK 66/22, it is being investigated whether the administration of the drug INT230-6 before surgery for breast cancer can increase the rate of pCR in the tumor and affected lymph nodes. The tolerability of INT230-6 as well as other factors such as response to treatment and the possibility of breast-conserving surgery are also being examined.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) poses significant challenges due to its aggressiveness, high relapse rates, and increased mortality. The Keynote-522 study revealed a 19.6% incidence of event-free survival (EFS) events in early-stage TNBC patients over 39 months. Achieving pathological complete response (pCR) and clearing positive lymph nodes are crucial prognostic factors.

The IMP INT230-6 is a combination of the chemotherapeutic agents cisplatin and vinblastine, along with a molecule that facilitates their distribution in tumor tissue. INT230-6, currently in clinical trials, has demonstrated the ability to induce up to 95% necrosis in T2 breast cancer tumors and it has been observed to stimulate systemic immune activation during the period between diagnosis and surgery. Moreover, promising results have been seen in seven refractory breast cancer patients, resulting in decreased Ki67 levels and a median overall survival of 12 months.

Completed and ongoing U.S. clinical trials including 91 patient a window-of-opportunity trial demonstrate the safety and early activity of INT230-6, both alone and with checkpoint inhibitors like pembrolizumab and ipilimumab, particularly in resistant cases.

Based on the positive outcomes, it will be assessed within this clinical trial the safety and early clinical activity of INT230-6 in early TNBC patients, addressing the high unmet medical need in this challenging subtype.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to country specific law and ICH GCP E6(R2) regulations before registration and prior to any trial specific procedures.
* Newly histologically diagnosed, previously untreated locally advanced non-metastatic TNBC as defined by the most recent American Society of Clinical Oncology (ASCO) / College of American Pathologist (CAP) guidelines .
* The following stages according to staging per American Joint Committee on Cancer (AJCC) for breast cancer staging criteria version 8 are included: cT1c (1.5-2cm) N1-3 M0 or cT2-4c N0-3 M0.
* Multifocal and multicentric primary tumors are allowed and the tumor with the most advanced T stage should be used to assess eligibility. If multifocal or multicentric disease TNBC needs to be confirmed for each focus.
* Measurable disease in the breast with at least one lesion with a diameter ≥ 1.5cm that is evaluable per RECIST v1.1, visible in ultrasound and injectable.
* Male or female subject Age ≥ 18 years.
* ECOG performance status 0-1
* Adequate bone marrow function (administration of G-CSF, EPO and/or blood transfusion within 14 days before registration is not allowed):

  * neutrophil count ≥ 1.5 x 109/L
  * platelet count ≥ 100 x 109/L
  * hemoglobin ≥ 90 g/L
* Adequate hepatic function:

  * total bilirubin ≤ 1.5 x ULN, or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN,
  * Albumin 30 ≥ g/L
  * Lactate Dehydrogenase (LDH) <2.5 ULN
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 50 ml/min/1.73 m2 (according to CKD-EPI formula)
* Adequate cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 50% as determined by echocardiography (ECHO)
* Adequate coagulation function:

  * INR ≤ 1.5 x ULN unless the patient is receiving anticoagulant therapy
  * aPTT ≤ 1.5 x ULN unless the patient is receiving anticoagulant therapy
  * If the patient is receiving anticoagulant therapy, the treating physician must determine that the anticoagulation can be stopped at least 24 hours prior to injection.
* Women of childbearing potential must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 7 months after the last dose of INT230-6 or 6 months after standard of care treatment. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential. (www.swissmedicinfo.ch).
* Men agree not to donate sperm or to father a child by using effective contraception during trial treatment and until 6 months after the last dose of INT230-6 or standard of care treatment (www.swissmedicinfo.ch).

Exclusion Criteria:

* Inflammatory Breast Cancer cT4d
* The following histological subtypes of TNBC are excluded: Classic adenoid cystic carcinoma, secretory carcinoma, low-grade adenosquamous carcinoma, tall cell carcinoma with reversed polarity, high-grade metaplastic
* History of invasive malignancy ≤3 years prior to signing informed consent (except treated basal cell or squamous cell skin cancer or in situ cervical cancer)
* Prior chemotherapy, targeted therapy, radiation therapy or anti-PD-L1 agent for previous breast cancer or Ductal Carcinoma in Situ (DCIS) on the same side.
* Concurrent bilateral breast cancer
* Concomitant treatment with any other experimental drug for recent breast cancer diagnosis in another clinical trial.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA II or IV; unstable angina pectoris, history of myocardial infarction and acute coronary syndrome requiring stenting/bypass surgery within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension.
* Known history of human immunodeficiency virus (HIV) or active chronic hepatitis C or hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
* Active autoimmune disease that required systemic treatment in past 2 years (e.g., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroid hormone replacement, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Known history of tuberculosis.
* Known history of allogeneic organ or stem cell transplant.
* Receipt of live attenuated vaccine (including yellow fever vaccine) within 30 days prior to registration.
* Diagnosis of immunodeficiency, concomitant or prior use of immunosuppressive medication within 7 days before registration, with the exceptions of local (intranasal, topical and inhaled) corticosteroids, or systemic corticosteroids which must not exceed 10 mg/day of prednisone or a dose equivalent corticosteroid, and the premedication for chemotherapy.
* Concomitant anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon), factor Xa inhibitors (e.g. rivaroxaban, apixaban), direct thrombin inhibitors (e.g. dabigatran) or platelet inhibitors/antiplatelet agents that cannot be stopped 24 hours before the administration of INT230-6. Aspirin (up to 300 mg/day) is allowed.
* Any concomitant drugs contraindicated for use with the trial drug according to the Investigator Brochure (IB) and the immuno-chemotherapy treatment according to the approved product information.
* Known hypersensitivity to trial drug or to any component of the trial drug or immuno-chemotherapy treatment.
* Incapacitated adults and any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) in the primary tumor (ypT0/Tis) and affected lymph nodes (ypN0). | At the date of tumor assessment after surgery, estimated at 29 to 32 weeks after treatment start for cohort A and at 27 to 30 weeks after treatment start for cohort B.
  The two following criteria need to be fulfilled for pCR:
  No invasive breast cancer in primary tumor (noninvasive breast residuals allowed) ypT0/Tis No invasive breast cancer in affected lymph nodes ypN0 The primary endpoint will be analyzed based on the resected patients set. The endpoint is evaluated according to the assessment of the local pathologist.

SECONDARY OUTCOMES:
pCR (invasive and in-situ, only invasive, respectively) in the breast | At the date of tumor assessment after surgery, estimated at 29 to 32 weeks after treatment start for cohort A and at 27 to 30 weeks after treatment start for cohort B.
  No invasive and no in situ breast cancer in primary tumor ypT0 No invasive breast cancer in affected lymph nodes ypN0 The endpoint will be analyzed based on the resected patients set. The endpoint is evaluated according to the assessment of the local pathologist.
pCR in lymph nodes | At the date of tumor assessment after surgery, estimated at 29 to 32 weeks after treatment start for cohort A and at 27 to 30 weeks after treatment start for cohort B.
  No invasive and no in situ breast cancer in primary tumor ypT0 No invasive breast cancer in affected lymph nodes ypN0 The endpoint will be analyzed based on the resected patients set. The endpoint is evaluated according to the assessment of the local pathologist.
Pattern of non pCR | At the date of tumor assessment after surgery, estimated at 29 to 32 weeks after treatment start for cohort A and at 27 to 30 weeks after treatment start for cohort B.
  Pattern in the remaining tumor is for example visible circle or tumor border, moon shaped residual tumor, islands of tumor in sea of necrosis, tumor streaks radiating from the main tumor into the surrounding tissue, single tumor cells (e.g. in lobulary tumor).
  This endpoint will be analyzed based on the subset of patients in the resected patients set who did not achieve pCR in the primary tumor (any invasive cancer in primary tumor).
Overall response according to RECIST v1.1 | At 1 to 4 weeks after last SOC treatment and before surgery, estimated at 27 to 30 weeks after treatment start for cohort A and at 25 to 28 weeks after treatment start for cohort B.
  Overall response (OR) is defined as complete response (CR) or partial response (PR) in the last pre-surgery tumor assessment compared with baseline MRI evaluated according to RECIST v1.1. In the subset of patients in cohort A additionally the change from baseline to the MRI between the 2nd injection and start of immunochemotherapy will be evaluated.
  The Criteria for RECIST v1.1. will be used with one modification: the injected lesion will still be measured/evaluated for this endpoint. Rationale: For a large proportion of the patients the injected lesion will be the only tumor lesion (cT2-4, cN0) or it will contain the majority of the tumor burden (in cN1 cases). Therefore, not evaluating this lesion would result in to many patients lost for this endpoint.
  This endpoint will be analyzed based on the FAS (Full Analysis Set).
Radiological tumor response using two perpendicular diameters | At 1 to 4 weeks after last SOC treatment and before surgery, estimated at 27 to 30 weeks after treatment start for cohort A and 25 to 28 weeks after treatment start for cohort B.
  Bidimensional assessment is only done for the largest (injected) primary tumor in the breast (not of satellite lesions and not of lymph nodes): we use the largest diameter measured in MRI and its perpendicular second diameter in the same MRI image. The two diameters are multiplied. Radiological tumor response in the last pre-surgery MRI is defined as follows:
  * CR: disappearance of the whole lesion
  * PR: > 50% decrease from baseline
  * PD: > 25% increase from baseline or appearance of new lesions in the breast This endpoint will be analyzed based on the FAS (Full Analysis Set).
Event free survival (EFS) | ): From the date of randomization until the date of the event of interest up to 3 years after surgery.
  EFS is defined as the time from randomization to any of the following events, whichever comes first:
  * Progression of disease that precludes surgery
  * Local or distant recurrence
  * Second primary malignancy (breast or other cancers). The following events are excluded: basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix lobular carcinoma in situ of the breast (LCIS), ductal carcinoma in situ of the breast (DCIS) and myeloplastic syndrome
  * Death due to any cause Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a subsequent treatment, if any.
  This endpoint will be analyzed based on the FAS.
Rate of breast conserving surgery (BCS) at the time of definitive surgery | At the date of surgery, estimated at 29 to 32 weeks after treatment start for cohort A and at 27 to 30 weeks after treatment start for cohort B.
  Proportion of patients with BCS at the time of definitive surgery. This endpoint will be analyzed based on the resected patients set.
Conversion of intention for mastectomy to BSC and axillary lymph node dissection (ALND) to sentinel lymph node dissection (SLND) or tailored axillary surgery (TAS) after treatment | At the date of pre-operative interdisciplinary tumor board assessment, estimated at 26 to 32 weeks after treatment start for cohort A and at 24 to 30 weeks after treatment start for cohort B
  This endpoint is defined as the change from intended mastectomy at baseline to BCS at time point of definitive surgery or from ALND to SLND or TAS.
  It will be analyzed based on the subgroup of the patients in the resected patients set for which mastectomy or ALND was foreseen at registration.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, Prof, Study Director — hoch Health Ostschweiz - Kantonsspital St. Gallen; Ursina Zürrer, MD, Study Chair — Kantonsspital Winterthur KSW
Locations (9):
- Switzerland (9):
  - Tumor Zentrum Aarau, Aarau
  - St. Claraspital, Basel
  - EOC - IOSI Ospedale regionale Bellinzona e valli - San Giovanni, Bellinzona
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Baselland, Liestal
  - HOCH Health Ostschweiz, Sankt Gallen
  - TBZO - Tumor- & Brustzentrum Ostschweiz, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich - Klinik für Gynäkologie, Zurich